CLINICAL TRIAL: NCT04358692
Title: Epicardial Measurement of Myocardial Stiffness on Beating Heart and Non-beating Heart During a Programmed Surgical Aortic Valve Replacement for Aortic Stenosis
Brief Title: Measurement of Myocardial Stiffness Using Elastometry in Patients With Aortic Stenosis
Acronym: ELASTOP-AS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/0254/HP
Record Dates: First submitted 2020-04-09; First posted 2020-04-24 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-04

CONDITIONS: Aortic Valve Stenosis
Keywords: Elastography; Myocardial stiffness; Surgical Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgical Aortic Valve Replacement (Experimental): Patients with aortic stenosis
  Interventions: Device: Aixplorer Mach30
- Reference (Other): Coronary bypass patients without hypertrophic left ventricular remodeling or sequelae of myocardial infarction
  Interventions: Device: Aixplorer Mach30

INTERVENTIONS:
Device: Aixplorer Mach30 — To measure myocardial stiffness by ShearWave elastography on not beating heart

SUMMARY:
Elastography is a new non-invasive medical technique for measuring the stiffness at a distance from a tissue. Recent advances in the development of elastography sequences for cardiac exploration suggest a more clinical approach to cardiac elastography. This study propose to compare myocardial stiffness of a group of coronary bypass patients without hypertrophic left ventricular remodeling or sequelae of myocardial infarction versus a group of patients who should benefit from a surgical aortic valve replacement for aortic stenosis.

The hypothesis is that the physiological adaptation to pressure overload constituted by aortic stenosis is responsible for a significant increase in myocardial stiffness compared to a reference group.

ELIGIBILITY:
Inclusion Criteria:

* Group I (aortic stenosis):

  1. Patient undergoing planned surgical aortic valve replacement (SAVR) for aortic stenosis (aortic valve area <1cm² or an aortic valve area index <0.6 cm² / m²);
* Group II: coronary bypass 2. Patient undergoing planned myocardial revascularization surgery (coronary bypass);
* Groups I and II 3. Patient over 18 years of age; 4. Patient having read and understood the information letter and having signed the consent form; 5. Patient affiliated or benefiting from a health insurance scheme

Exclusion Criteria:

* Group II: coronary bypass

  1. Ratio in TM mode of the wall thickness over the radius of the left ventricle (h / r [0.45]) confirmed by the TTE;
  2. Scar of myocardial infarction defined by an ECG anomaly and / or hypo-akinesia on TTE, and / or a late enhancement in MRI;
  3. Acute coronary syndrome less than 3 months old;
  4. Significant aortic stenosis (Vmax> 1.5 m / s);
  5. Anomaly of segmental kinetics;
  6. Presence of left ventricular hypertrophy
* Groups I and II 7. Mitral valve disease (> 1/4 confirmed by TTE); 8. Aortic insufficiency (> 1/4 confirmed by TTE); 9. Left ventricle ejection fraction (LVEF) <50% confirmed by TTE; 10. Hospitalization for heart failure less than 3 months old; 11. Urgent surgery; 12. Infiltrative heart disease; 13. Hostile pericardium defined by a history of mediastinal radiotherapy, tamponade or complicated pericarditis; 14. Decompensated or severe arterial hypertension. 15. Functional inability to walk preventing the performance of the walk test; 16. Proven pregnant woman (positive urine pregnancy test) or breastfeeding or absence of effective contraception (as defined by the WHO) or postmenopausal woman without confirmation diagnosis obtained (amenorrhea not medically induced for at least 12 months before the initiation visit) ; 17. Person deprived of their liberty by an administrative or judicial decision or person placed under the protection of justice / guardianship or curatorship 18. History of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participating in the protocol or preventing him from giving his informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
to compare myocardial stiffness by ShearWave elastography on not beating heart in two groups of patients referred for surgery | Day 1
  The main outcome measure is evaluated by ShearWave elastography with the measurement of Young modulus on non-beating heart

SECONDARY OUTCOMES:
To compare the diastolic myocardial stiffness of the beating heart with the myocardial stiffness of the non-beating heart | Day 1
  This outcome measure is evaluated by ShearWave elastography with the measurement of Young modulus on non-beating heart
To compare epicardial and trans-thoracic diastolic myocardial stiffness | Day 1
  This outcome measure is evaluated by elastography using the measurement of Young modulus in epicardial (using the linear probe) and transthoracic (using the scanning probe).
Correlation between the diastolic myocardial stiffness of the beating heart and the non-beating heart with conventional diastolic indices | Day 1
  This outcome measure is evaluated:
  1. by ShearWave elastography with the measurement of Young modulus on non-beating heart
  2. by conventional ultrasound criteria (peak e', peak E, volume of the left atrium calculated by simpson biplanes, maximum velocity of tricuspid insufficiency).
Correlation between the diastolic myocardial stiffness of the beating heart and the non-beating heart with heart failure parameters | Day 1
  This outcome measure is evaluated:
  1. by ShearWave elastography with the measurement of Young modulus on non-beating heart
  2. by heart failure parameters defined by NYHA class, the walking test and the BNP assay
Correlation between the diastolic myocardial stiffness of the beating heart and the non-beating heart with left ventricular mass indexed to the body surface | Day 1
  This outcome measure is evaluated:
  1. by ShearWave elastography with the measurement of Young modulus on non-beating heart
  2. by LV mass indexed to the body surface calculated by the cardiac mass measuring by ultrasound indexed to the body surface
Correlation between the diastolic myocardial stiffness of the beating heart and the non-beating heart and the prognosis | 1 year
  This outcome measure is evaluated:
  1. by ShearWave elastography with the measurement of Young modulus on non-beating heart
  2. by a combined index combining all rehospitalization for heart failure, increase in heart failure treatment and cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Eric Saloux, MD, Study Director — University Hospital, Caen
Locations (2):
- France (2):
  - CHU Caen, Caen
  - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No